CLINICAL TRIAL: NCT07277634
Title: Cultural Adaptation and Validity-Reliability of Attitude Scales Toward Artificial Intelligence in Turkish: A Psychometric Study on Physical Therapy Patients
Brief Title: Cultural Adaptation of Attitude Scales Towards Artificial Intelligence Into Turkish
Status: Not yet recruiting | Type: Observational
Sponsor: Barış SEVEN (Other)
Responsible Party: Sponsor-Investigator, Barış SEVEN, Ph.D, Gazi University
Organization: Gazi University (Other)
Other Study IDs: 10
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Physical Therapy Patient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physical therapy patients

SUMMARY:
The rapid proliferation of artificial intelligence (AI) applications in healthcare has led to significant transformations, particularly in applications such as patient management, treatment planning, clinical decision support systems, and remote rehabilitation. Ensuring that this transformation is effective and safe requires the reliable measurement of patients' perceptions and attitudes toward AI-based health technologies. However, the existing literature does not include any scales developed to measure patients' attitudes toward AI that have been adapted to Turkish society. This situation complicates both the assessment of acceptance of AI in clinical applications and the sound execution of scientific research in this field.

This research aims to culturally adapt the internationally developed ATTARI-12 (Attitudes Toward Artificial Intelligence-12) and ATTARI-WHE (Artificial Intelligence in Work, Health and Everyday Life) scales into Turkish and to evaluate their construct validity and reliability. The study is methodological in design and will be conducted at the Faculty of Health Sciences, Izmir Katip Celebi University, between January 2026 and January 2027, following approval by the ethics committee. The cultural adaptation method proposed by Beaton and colleagues, which includes forward translation, back translation, expert panel, and content validity stages, will be applied during the scale adaptation process; then, the understandability of the items will be tested with a pilot application. The sample will consist of at least 200 physical therapy patients, and convergent validity, construct validity using confirmatory factor analysis, and reliability using Cronbach's alpha and test-retest methods will be evaluated.

The project will be carried out according to a structured schedule consisting of project management, translation process, pilot application, data collection, and analysis stages. All measurements will be performed after obtaining ethical committee approval.

The results of this study will contribute to the literature by providing patient-specific, valid, and reliable measurement tools that can be used to scientifically evaluate patients' attitudes toward AI in Turkey. These scales are expected to have a widespread impact in national research, in the evaluation of clinical decision support systems, and in strategies aimed at increasing the acceptance of AI-based health technologies.

DETAILED DESCRIPTION:
This is a Cultural Adaptation and Validity-Reliability study

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing active treatment in the Physical Therapy and rehabilitation unit.
* Being cognitively able to answer the questionnaire.

Exclusion Criteria:

* Severe communication or cognitive impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing active treatment in the Physical Therapy and rehabilitation unit
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ATTARI-12 (Attitudes Toward Artificial Intelligence-12) and ATTARI-WHE (Artificial Intelligence in Work, Health and Everyday Life) Scales | From January 2026 to January 2027